CLINICAL TRIAL: NCT00779064
Title: BAY59-7939, Japanese Phase II in Atrial FibrillationTrial Status
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11390
Record Dates: First submitted 2008-10-17; First posted 2008-10-24 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)
- Arm 2 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (BAY59-7939) — 10mg BID, Semi-sequential, dose escalation.
  Arms: Arm 1
Drug: Rivaroxaban (BAY59-7939) — 20mg BID, Semi-sequential, dose escalation.
  Arms: Arm 2

SUMMARY:
This is a clinical study investigating pharmacokinetics, pharmacodynamic effects and safety of BAY 59-7939 in patients with atrial fibrillation (originally described in Japanese).

ELIGIBILITY:
Inclusion Criteria:

* 20 years or older
* Japanese male or female
* Non- valvular atrial fibrillation documented by ECG
* Patients aged 60 years and older or with a risk of stroke

Exclusion Criteria:

* Prior stroke and TIA
* Patients in whom anticoagulants are contraindicated

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-07; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) CL/f, AUC, Cmax, Pharmacodynamics (PD), Factor Xa activity, PT, PT-INR, aPTT and HEPTEST(R) | Day 14 and 28

SECONDARY OUTCOMES:
Each category of bleeding events and adverse event | Throughout treatment and followup period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- Japan (9):
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Kurume, Fukuoka
  - Kitahiroshima, Hokkaido
  - Amagasaki, Hyōgo
  - Kawachi-Nagano, Osaka
  - Osaka, Osaka
  - Suita, Osaka